CLINICAL TRIAL: NCT05736679
Title: EaveTubes for Control of Vector Borne Diseases in Côte d'Ivoire
Brief Title: EaveTubes for Vector Control
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Notre Dame (Other)
Collaborators: Institut Pierre Richet (Other Government); In2Care (Unknown)
Responsible Party: Principal Investigator, John Grieco, Research Professor, University of Notre Dame
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 22-10-7454
Record Dates: First submitted 2023-02-10; First posted 2023-02-21 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Malaria
Keywords: EaveTubes; Housing; Malaria control; LLINs; Cost-effectiveness; Malaria; Vector-borne diseases; Mosquito vectors; Incidence
MeSH Terms: conditions — Malaria; Vector Borne Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Given the nature of the intervention, it is impossible to conduct this study in a fully blinded manner but those parts of the data collection that can be blinded will be. Observer bias will be reduced where feasible. All laboratory work will be blinded. Mosquito collector bias will be reduced by using standard light traps which do not rely on the ability of the fieldworker to collect specimens. Trap catches will not be examined and analyzed by those who collected them but by different technicians who will not know the trap location. We will use codes to identify any clinical samples. Electronic records will not carry the name of the research participants, only an alphanumeric code. Primary analysis by the project statistician will be conducted on blinded data (e.g. arms designated as treatment A & B or something similar). Datasets will only be unblinded once they have been locked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- In2Care EaveTube (Experimental): EaveTube installation with deltamethrin treated netting; in addition to standard of care (standard pyrethroid-only bednets)
  Interventions: Device: In2Care EaveTube
- Control (No Intervention): Standard of care (standard pyrethroid-only bednets)

INTERVENTIONS:
Device: In2Care EaveTube — In2Care® EaveTubes (ETs) comprise 15 cm diameter, 20 cm long ventilation tubes with removable netting inserts that are placed in the wall under the roof of houses where they attract malaria mosquitoes at night, block them from entering the house, and contaminate them with a lethal dose of insecticide. In2Care® ET netting inserts have an electrostatically charged coating treated with bio-actives in powder form, which kills insecticide-resistant mosquitoes through high active ingredient dose transfer.
  Arms: In2Care EaveTube

SUMMARY:
The goal of this clinical trial is to test whether In2Care EaveTubes (ETs) as a stand-alone tool can reduce malaria in an area where transmission is driven by insecticide-resistant Anopheles gambiae. Children who live in homes with ETs will be monitored for malaria infection and compared to children living in homes without ETs in Côte d'Ivoire where there is universal coverage of long lasting insecticide nets and pyrethroid resistance is high.

DETAILED DESCRIPTION:
In2Care EaveTubes (ETs) are an inexpensive, new vector control product under World Health Organization (WHO) evaluation informed by mosquito ecology to efficiently target malaria vectors. By installing ETs in the walls of the house at eave level that funnel the natural airflow, mosquitoes are drawn in by the same heat and odor cues that typically attract them through the eaves. Once inside an ET, mosquitoes come into contact with insecticide-treated netting placed inside the ET.

The aim of this study is to test whether ETs as stand-alone tool have an effect on the epidemiology of malaria in villages where houses have been modified with the ET intervention. This prospective 2-arm cluster randomized control trial based on a WHO Vector Control Advisory Group approved protocol will include 17 intervention clusters and 17 control clusters. Both arms will have pyrethroid-treated bednets. Based on the population census, 55 households per cluster with eligible children will be randomly selected for recruitment into the active detection cohorts. In the intervention arm, we will enroll eligible children who reside in ET-treated houses. In the control arm, we will enroll children residing in villages without ET-treated houses. The intervention and control cohorts will be followed for 4 months for baseline covariate measurements and 24 months of a clinical follow up period. During case detection visits, blood samples will be taken from all febrile children and tested for malaria infection with rapid diagnostic tests. To assess the impact of the ET on mosquito density, entomological measurements will be conducted monthly in 20 clusters (10 ET, 10 Control) in 10 randomly selected households per cluster. To estimate the infectiousness of malaria vectors, sporozoite rates will be measured in subsets of the collected mosquito samples.

ELIGIBILITY:
Village Level Inclusion Criteria:

* ≥ 80% of Households (HHs) must be suitable for EaveTube(ET) installation.
* ≥70% of HHs willing to have ETs installed.
* No participation in the previous Screening + ETs cluster randomized control trial (cRCT).
* Received standard pyrethroid-only long lasting insecticide nets(LLINs) (Permanet 2.0).
* 100-300 HHs per village.
* ≥2 km apart from another village.

Village Level Exclusion Criteria:

* < 80% of HHs suitable for ET installation.
* <70% of HHs willing to have ETs installed.
* Villages being treated by indoor residual spray (IRS) and/or new generation bed net campaigns.
* Participation in previous Screening + ET cRCT.
* <100 and >300 households per village.
* <2 km from another village.

Household Level Inclusion Criteria

* HHs must be suitable for ET installation.
* Provision of consent from heads of HH.

Household Level Exclusion Criteria

* HH not suitable for ET installation (e.g. houses with poor quality thatch roofing or very large eaves or wall gaps, houses in substantial disrepair, unfinished houses under construction, poorly constructed houses, ).
* No provision of consent from heads of HH.

Individual Level Inclusion Criteria

* Children aged ≥ 6 months to < 8 years old at time of enrollment (so all participants are under 10 years old for the duration of clinical follow-up).
* Provision of written, informed consent by parents/care givers.
* Children must reside in villages enrolled in the study and in ETs-treated HHs.
* Hemoglobin at baseline of >7 mg/dL.

Individual Level Exclusion Criteria

* Children aged < 6 months or ≥ 8 years old at time of enrollment.
* No provision of written, informed consent by parents/care givers for child participation.
* Expected to be non-resident during a significant part of the transmission season.
* Hemoglobin at baseline of ≤7 mg/dL, have a known chronic disease, or who have signs of clinical decompensation.
* Participation in another clinical trial investigating a drug, vaccine, medical device or procedure.

Ages: 6 Months to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1870 (Estimated)
Dates: Start 2023-03-23 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of malaria infection | 24 months
  Measured by active infection and clinical malaria case detection in cohorts of 55 children (between 6 months and 10 years old) per cluster, 17 clusters per arm on a biweekly basis in peak transmission season and monthly basis in low transmission season.

SECONDARY OUTCOMES:
Clinical malaria incidence | 24 months
  Measured in children between 6 months to 10 years old living in the study cohorts using passive case detection via the existing community health workers and health centers.
Malaria parasitemia | 24 months
  Measured in children between 6 months to 10 years old in the cohorts of 55 children.
Prevalence of moderate (defined as 7 - 9.9 g/dL hemoglobin) to severe anemia (<7 g/dL hemoglobin) | 24 months
  Measured in children under 5 years of age in the cohorts of 55 children four times: at the start and end of the rainy season (April and November respectively) of Year 1 and Year 2.
Mean numbers of female malaria mosquitoes (An. gambiae s.l., An funestus s.l.) captured in study houses | 24 months
  Measured by CDC light traps in 20 clusters, 10 houses per cluster on a monthly basis.
Malaria parasite sporozoite rate | 24 months
  Assessed in 10% of all anophelines captured by CDC light trap.
Entomological Inoculation Rates | 24 months
  Measured in each study arm as the product of the anopheline vector density and sporozoite rate.

OTHER OUTCOMES:
Cost-effectiveness of EaveTubes compared to the previously applies Screening + EaveTubes intervention, and compared to other vector control interventions such as LLINs and IRS. | 24 months
  Cost modelling will assess cost-effectiveness of EaveTubes compared to the previously applies Screening + EaveTubes intervention, and compared to other vector control interventions such as long lasting insecticide nets and indoor residual spray.
User acceptance of EaveTubes | 24 months
  Assessments of willingness to participate and adoption of EaveTubes at the end of the study period through questionnaires and willing to pay surveys.

CONTACTS AND LOCATIONS:
Overall Officials: John P Grieco, PhD, Principal Investigator — University of Notre Dame
Locations (1):
- Institut Pierre Richet, Bouaké, Côte d’Ivoire

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andriessen R, Snetselaar J, Suer RA, Osinga AJ, Deschietere J, Lyimo IN, Mnyone LL, Brooke BD, Ranson H, Knols BG, Farenhorst M. Electrostatic coating enhances bioavailability of insecticides and breaks pyrethroid resistance in mosquitoes. Proc Natl Acad Sci U S A. 2015 Sep 29;112(39):12081-6. doi: 10.1073/pnas.1510801112. Epub 2015 Aug 31. PMID 26324912
- [Background] Barreaux AMG, Brou N, Koffi AA, N'Guessan R, Oumbouke WA, Tia IZ, Thomas MB. Semi-field studies to better understand the impact of eave tubes on mosquito mortality and behaviour. Malar J. 2018 Aug 22;17(1):306. doi: 10.1186/s12936-018-2457-4. PMID 30134907
- [Background] Barreaux AMG, Oumbouke WA, Tia IZ, Brou N, Koffi AA, N'guessan R, Thomas MB. Semi-field evaluation of the cumulative effects of a "Lethal House Lure" on malaria mosquito mortality. Malar J. 2019 Aug 30;18(1):298. doi: 10.1186/s12936-019-2936-2. PMID 31470873
- [Background] Bhatt S, Weiss DJ, Cameron E, Bisanzio D, Mappin B, Dalrymple U, Battle K, Moyes CL, Henry A, Eckhoff PA, Wenger EA, Briet O, Penny MA, Smith TA, Bennett A, Yukich J, Eisele TP, Griffin JT, Fergus CA, Lynch M, Lindgren F, Cohen JM, Murray CLJ, Smith DL, Hay SI, Cibulskis RE, Gething PW. The effect of malaria control on Plasmodium falciparum in Africa between 2000 and 2015. Nature. 2015 Oct 8;526(7572):207-211. doi: 10.1038/nature15535. Epub 2015 Sep 16. PMID 26375008
- [Background] Bradley J, Rehman AM, Schwabe C, Vargas D, Monti F, Ela C, Riloha M, Kleinschmidt I. Reduced prevalence of malaria infection in children living in houses with window screening or closed eaves on Bioko Island, equatorial Guinea. PLoS One. 2013 Nov 13;8(11):e80626. doi: 10.1371/journal.pone.0080626. eCollection 2013. PMID 24236191
- [Background] Carey JR, Muller HG, Wang JL, Papadopoulos NT, Diamantidis A, Koulousis NA. Graphical and demographic synopsis of the captive cohort method for estimating population age structure in the wild. Exp Gerontol. 2012 Oct;47(10):787-91. doi: 10.1016/j.exger.2012.06.012. Epub 2012 Jul 7. PMID 22776134
- [Background] Hayes RJ, Bennett S. Simple sample size calculation for cluster-randomized trials. Int J Epidemiol. 1999 Apr;28(2):319-26. doi: 10.1093/ije/28.2.319. PMID 10342698
- [Background] Kirby MJ, Ameh D, Bottomley C, Green C, Jawara M, Milligan PJ, Snell PC, Conway DJ, Lindsay SW. Effect of two different house screening interventions on exposure to malaria vectors and on anaemia in children in The Gambia: a randomised controlled trial. Lancet. 2009 Sep 19;374(9694):998-1009. doi: 10.1016/S0140-6736(09)60871-0. Epub 2009 Sep 3. PMID 19732949
- [Background] Koffi AA, Ahoua Alou LP, Adja MA, Chandre F, Pennetier C. Insecticide resistance status of Anopheles gambiae s.s population from M'Be: a WHOPES-labelled experimental hut station, 10 years after the political crisis in Cote d'Ivoire. Malar J. 2013 May 4;12:151. doi: 10.1186/1475-2875-12-151. PMID 23641777
- [Background] Koffi AA, Ahoua Alou LP, Kabran JP, N'Guessan R, Pennetier C. Re-visiting insecticide resistance status in Anopheles gambiae from Cote d'Ivoire: a nation-wide informative survey. PLoS One. 2013 Dec 16;8(12):e82387. doi: 10.1371/journal.pone.0082387. eCollection 2013. PMID 24358177
- [Background] Krajacich BJ, Slade JR, Mulligan RF, LaBrecque B, Alout H, Grubaugh ND, Meyers JI, Fakoli LS 3rd, Bolay FK, Brackney DE, Burton TA, Seaman JA, Diclaro JW 2nd, Dabire RK, Foy BD. Sampling host-seeking anthropophilic mosquito vectors in west Africa: comparisons of an active human-baited tent-trap against gold standard methods. Am J Trop Med Hyg. 2015 Feb;92(2):415-21. doi: 10.4269/ajtmh.14-0303. Epub 2014 Nov 24. PMID 25422393
- [Background] Lengeler C. Insecticide-treated bednets and curtains for preventing malaria. Cochrane Database Syst Rev. 2000;(2):CD000363. doi: 10.1002/14651858.CD000363. PMID 10796535
- [Background] Lindsay SW, Snow RW. The trouble with eaves; house entry by vectors of malaria. Trans R Soc Trop Med Hyg. 1988;82(4):645-6. doi: 10.1016/0035-9203(88)90546-9. No abstract available. PMID 3256125
- [Background] Lwetoijera DW, Kiware SS, Mageni ZD, Dongus S, Harris C, Devine GJ, Majambere S. A need for better housing to further reduce indoor malaria transmission in areas with high bed net coverage. Parasit Vectors. 2013 Mar 7;6:57. doi: 10.1186/1756-3305-6-57. PMID 23497471
- [Background] Oumbouke WA, Tia IZ, Barreaux AMG, Koffi AA, Sternberg ED, Thomas MB, N'Guessan R. Screening and field performance of powder-formulated insecticides on eave tube inserts against pyrethroid resistant Anopheles gambiae s.l.: an investigation into 'actives' prior to a randomized controlled trial in Cote d'Ivoire. Malar J. 2018 Oct 22;17(1):374. doi: 10.1186/s12936-018-2517-9. PMID 30348154
- [Background] Oumbouke WA, Pignatelli P, Barreaux AMG, Tia IZ, Koffi AA, Ahoua Alou LP, Sternberg ED, Thomas MB, Weetman D, N'Guessan R. Fine scale spatial investigation of multiple insecticide resistance and underlying target-site and metabolic mechanisms in Anopheles gambiae in central Cote d'Ivoire. Sci Rep. 2020 Sep 15;10(1):15066. doi: 10.1038/s41598-020-71933-8. PMID 32934291
- [Background] Pinder M, Conteh L, Jeffries D, Jones C, Knudsen J, Kandeh B, Jawara M, Sicuri E, D'Alessandro U, Lindsay SW. The RooPfs study to assess whether improved housing provides additional protection against clinical malaria over current best practice in The Gambia: study protocol for a randomized controlled study and ancillary studies. Trials. 2016 Jun 3;17(1):275. doi: 10.1186/s13063-016-1400-7. PMID 27255167
- [Background] Snetselaar J, Njiru BN, Gachie B, Owigo P, Andriessen R, Glunt K, Osinga AJ, Mutunga J, Farenhorst M, Knols BGJ. Eave tubes for malaria control in Africa: prototyping and evaluation against Anopheles gambiae s.s. and Anopheles arabiensis under semi-field conditions in western Kenya. Malar J. 2017 Jul 4;16(1):276. doi: 10.1186/s12936-017-1926-5. PMID 28778169
- [Background] Sternberg ED, Ng'habi KR, Lyimo IN, Kessy ST, Farenhorst M, Thomas MB, Knols BG, Mnyone LL. Eave tubes for malaria control in Africa: initial development and semi-field evaluations in Tanzania. Malar J. 2016 Sep 1;15(1):447. doi: 10.1186/s12936-016-1499-8. PMID 27586055
- [Background] Sternberg ED, Cook J, Alou LPA, Assi SB, Koffi AA, Doudou DT, Aoura CJ, Wolie RZ, Oumbouke WA, Worrall E, Kleinschmidt I, N'Guessan R, Thomas MB. Impact and cost-effectiveness of a lethal house lure against malaria transmission in central Cote d'Ivoire: a two-arm, cluster-randomised controlled trial. Lancet. 2021 Feb 27;397(10276):805-815. doi: 10.1016/S0140-6736(21)00250-6. PMID 33640067
- [Background] Tusting LS, Ippolito MM, Willey BA, Kleinschmidt I, Dorsey G, Gosling RD, Lindsay SW. The evidence for improving housing to reduce malaria: a systematic review and meta-analysis. Malar J. 2015 Jun 9;14:209. doi: 10.1186/s12936-015-0724-1. PMID 26055986
- [Background] Tusting LS, Bottomley C, Gibson H, Kleinschmidt I, Tatem AJ, Lindsay SW, Gething PW. Housing Improvements and Malaria Risk in Sub-Saharan Africa: A Multi-Country Analysis of Survey Data. PLoS Med. 2017 Feb 21;14(2):e1002234. doi: 10.1371/journal.pmed.1002234. eCollection 2017 Feb. PMID 28222094
- [Background] Wanzirah H, Tusting LS, Arinaitwe E, Katureebe A, Maxwell K, Rek J, Bottomley C, Staedke SG, Kamya M, Dorsey G, Lindsay SW. Mind the gap: house structure and the risk of malaria in Uganda. PLoS One. 2015 Jan 30;10(1):e0117396. doi: 10.1371/journal.pone.0117396. eCollection 2015. PMID 25635688
- [Background] Sperling S, Cordel M, Gordon S, Knols BGJ, Rose A. Eave tubes for malaria control in Africa: Videographic observations of mosquito behaviour in Tanzania with a simple and rugged video surveillance system. Malariaworld J. 2017 Jul 1;8:9. eCollection 2017. PMID 34532232
- [Background] Waite JL, Lynch PA, Thomas MB. Eave tubes for malaria control in Africa: a modelling assessment of potential impact on transmission. Malar J. 2016 Sep 2;15(1):449. doi: 10.1186/s12936-016-1505-1. PMID 27590602
- [Derived] N'Guessan R, Assi SB, Koffi A, Ahoua Alou PL, Mian A, Achee NL, Fustec B, Grieco JP, Liu F, Kumar S, Noffsinger M, Hudson A, Mohlmann TWR, Farenhorst M. EaveTubes for control of vector-borne diseases in Cote d'Ivoire: study protocol for a cluster randomized controlled trial. Trials. 2023 Nov 2;24(1):704. doi: 10.1186/s13063-023-07639-9. PMID 37919815
- See also: World Health Organization - Global plan for insecticide resistance management in malaria vectors. — https://www.who.int/publications/i/item/WHO-HTM-GMP-2012.5
- See also: World Health Organization, 2019 - Eleventh meeting of the WHO Vector Control Advisory Group — https://www.who.int/publications/i/item/9789240000759
- See also: MacDonald, M. (2015) Landscape of new vector control products. VectorWorks. — https://www.up.ac.za/media/shared/236/ZP_Files/VectorWorks/vector-control-landscape-2015_2.zp73113.pdf
- See also: Anderson L., Simpson D., Stephens M. (2014) Effective Malaria Control Through Durable Housing Improvements: Can we learn new strategies from past experience? Habitat Humanity International Global Programs Department — https://citeseerx.ist.psu.edu/document?repid=rep1&type=pdf&doi=4b41af5f2ae4722759692bee186c91857b91d663
- See also: Uganda Housing Modification Study (UHMS) — https://clinicaltrials.gov/ct2/show/NCT04622241?term=eave+tube&draw=2&rank=1